CLINICAL TRIAL: NCT01543321
Title: Study of Efficacy and Acceptability of Tetrabenazine in the Late Dyskinetic Syndrome With Neuroleptics: A Randomized, Parallel Group, Double-blind Placebo Controlled Multicentre Trial
Brief Title: Xenazine in Late Dyskinetic Syndrome With Neuroleptics
Acronym: Xeladys
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI11-PR-KRYSTKOWIAK; 2011-004211-23 (EudraCT Number)
Record Dates: First submitted 2012-02-22; First posted 2012-03-02 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tardive Dyskinesia
Keywords: tetrabenazine; movement disorders; tardive disorders
MeSH Terms: conditions — Tardive Dyskinesia; Movement Disorders | interventions — Tetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetrabenazine group (Experimental): Tetrabenazine is a drug that is administered orally. This is 25 mg tablets, divisible into 2.
  Interventions: Drug: Tetrabenazine
- Plagebo group (Placebo Comparator): Patients will receive a buccal tablet identical to the experimental product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrabenazine — Treatment with tetrabenazine consists in:
  * 5-week titration to a maximum dose of 200 mg / day
  * 5 weeks at stable dose
  * 2 weeks in wash-out
  The treatment will be blinded for patients and investigators
  Other Names: Xenazine (tetrabenazine)
  Arms: Tetrabenazine group
Drug: Placebo — Treatment with placebo consists in:
  * 5-week titration to a maximum dose of 200 mg / day
  * 5 weeks at stable dose
  * 2 weeks in wash-out
  The treatment will be blinded for patients and investigators
  Arms: Plagebo group

SUMMARY:
Late dyskinetic syndrome with neuroleptics, or tardive dyskinesia, is the appearance of abnormal involuntary movements (AIM) in patients treated with antipsychotics for at least three months. This important public health issue arises for 15-20% of patients treated with neuroleptics, the most prescribed psychotropic drugs in mental disorders in France, and seriously impacts the patients' quality of life. In over 50% of cases, it is irreversible-that is to say that he will persist despite discontinuation of the offending drug.

Risk factors have been described: the age and female gender are established, a higher dosage of antipsychotic, a long-term treatment, a psychiatric condition other than schizophrenia are likely risk factors, intermittent treatment, previous acute dyskinesia, neuroleptics or powerful, longer term use of corrective treatments including anticholinergics are still discussed.

Apart from preventive treatment, which consists in using antipsychotics as being coerced, support is disappointing: the etiological treatment, which is to stop the offending antipsychotic, is effective only in less than 50% of cases, the syndrome is most often late irreversible. Must still have the possibility to interrupt the treatment, which is usually impossible in the risk of decompensation of the mental illness for which the neuroleptic was prescribed. Remains symptomatic treatment: functional neurosurgery is only for extreme cases, because it is not without risk, in terms of morbidity and mortality. So it's the medication that is most often offered: many drugs have been proposed, a direct result of the multiplicity of neurotransmitter systems implicated.

However, in the vast majority of cases, this approach is disappointing not to say ineffective. The only exception is the tetrabenazine, marketed under the name of Xenazine®. Empirically, neurologists specializing in pathology of the movement are almost unanimous: its efficiency is very good, with good tolerance. Some preliminary studies have reinforced this impression. However, their level of evidence remains low and that is why the investigators propose to implement a prospective multicenter clinical trial, double-blind with placebo which will include two groups of 27 patients.

DETAILED DESCRIPTION:
Tetrabenazine is classified as a central monoamine depleting agent. In vitro studies have shown that it is an inhibitor of the vesicular monamine transporter 2 (VMAT2), resulting in synaptic dopamine depletion. This effect explains the reduction of hyperkinetic movement disorders.

Although tetrabenazine enjoys a reputation of very good efficacy in tardive syndromes, with good tolerance, it is still yet to empiricism because studies are few andf most importantly, of low level of evidence according the criteria of Evidence Based Medicine.

This is a randomized, multicenter, parallel group, double-blind placebo (tetrabenazine/placebo: 1/1), in two comparative conditions before and after 10 weeks of treatment with tetrabenazine (5-week titration to a maximum dose of 200 mg/day and 5 weeks at stable dose).

Study enrollment is proposed to patients fulfilling inclusion criteria.

The study should process as follows:

1. Patients give their informed consent for participation after presentation of the study by the investigator.
2. Visit V0: Given the patient's signed consent, global clinical examination, blood sampling, vital signs (weight, height, arterial tension, ECG are performed as well as a neurological examination (MMS). For women in childbearing potential, a urinary pregnancy test will be realized. It is noteworthy that a psychiatric consultation dating less than one month is required.
3. Visit V1: patient is randomized in one of the two arms: tetrabenazine or placebo. Some tests are performed at baseline:

   * Neurologic: ESRS, AIMS, CGI, UPDRSIII, MMS;
   * Quality of life auto-questionnaires: SF36, Epworth; The treatment is prescribed following a titration phase during 5 weeks, a stable dose during 5 weeks, and a wash-out period during 2 weeks.
4. At V2 (1 week after V1), V3 (3 weeks after V1) and V5 (7 weeks after V1): global clinical examination is performed and prescription observance is checked.
5. At V4 (5 weeks after V1), V6 (10 weeks after V1) and V7 (12 weeks after V1): neurological (ESRS, AIMS, CGI, UPDRSIII, auto questionnaire SF36, Epworth, neuropsychological examination (MADRS), psychiatric examination (only at V6), vital signs and prescription observance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age over 18) or adult under judicial protection (tutor or curator).
2. Patient with late dyskinetic syndrome with neuroleptics yielding functional disability and/or impact in every day's life, according to the investigator, and/or the patient and/or the patient's family.
3. Patient with persistent late dyskinetic syndrome, even if the neuroleptic has been stopped for more than 6 months or patient with late dyskinetic syndrome under neuroleptic treatment unchanged for at least 3 months and which would a priori not need any dose variation during the study time.
4. MADRS < 18
5. QTc < 450 ms for men and < 470 for women.

Exclusion Criteria:

1. Lack of social insurance
2. Neuroleptic treatment less than 3 months
3. Insanity according to the DSM IV and MMS < 24
4. Predominant akathisia
5. Psychiatric disease not stabilized for more than 6 months and/or which could require a neuroleptic treatment adaptation during study time.
6. Pregnancy and lactating
7. Women in genital activity without efficient contraception method (IUD or estrogen-progestin pill)
8. Hypersensitivity to tetrabenazine
9. Renal failure
10. Drugs: Non-selective MAOIs, dopaminergic (or other antiparkinsonian)
11. Other severe pathology
12. Patient non compliant to protocol, at the investigator's appreciation
13. Simultaneous participation to other clinical trial
14. Congenital galactosemia, glucose malabsorption or lactase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes in ESRS: Extrapyramidal Symptoms Rating Scale | 10 weeks after randomization
  Changes in ESRS from Baseline and V6 (10 weeks after randomization) are assessed at the end of the 10 weeks of treatment.

SECONDARY OUTCOMES:
Changes in Sub-score ESRS-II | At baseline (V1), V4 (7 weeks after V1), V6 (10 weeks after V1) and V7 (14 weeks after V1)
  ESRS-II is calculated as the ESRS total score minus ESRS sub-part II (worst score=0, best score=158).
  The choice of this sub-score is justified because of the possibility of improving the total ESRS can be masked by the induction of parkinsonian syndrome represented by part II of the ESRS that we chose to subtract in order to achieve the ESRS 2.
CGI amelioration | At baseline (V1), V4 (7 weeks after V1), V6 (10 weeks after V1) and V7 (14 weeks after V1)
  Clinical Global Impression is an ordinal scale in eight categories: unevaluated = 0; much worsened = 7
Tolerance | within the 14 weeks of the patients' participation
  Tolerance includes:
  * neurological consultation
  * global clinical examination: ECG (QT), BP, pulse, orthostatic hypotension, weight
Changes in Quality of life | At baseline (V1), V4 (7 weeks after V1), V6 (10 weeks after V1) and V7 (14 weeks after V1)
  Quality of life will be investigated with the SF36 questionnaire.
AIMS improvement | At baseline (V1), V4 (7 weeks after V1), V6 (10 weeks after V1) and V7 (14 weeks after V1)
  Expected reduction of dyskinesia during the study will be investigated with the Abnormal Involuntary Movement Scale (AIMS).
Changes in intermediate ESRS and post-treatment ESRS | 7 weeks after randomization and 14 weeks after randomization
  Changes in ESRS are assessed between baseline and the end of the titration period (7 weeks after randomization) and after the wash-out period (14 weeks after randomization).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krystkowiak, MD-PhD, Principal Investigator — University Hopsital of Amiens
Locations (19):
- France (19):
  - CHU Amiens, Amiens, Picardie
  - CH Aix en Provence, Aix-en-Provence
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CH des Charpennes, Lyon
  - AP-HM Hopital de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHRU de Nimes, Nîmes
  - CHU Saint Antoine, Paris
  - CHU Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

REFERENCES:
- [Result] Neurologies • Janvier 2012 • vol. 15 • numéro 144 page 35 http://association.gens.free.fr/NEUROLOGIA/Revues%20Neuro%20Articles/EXTRAPYRAMIDAL/$syndrome%20tardif%20aux%20neuroleptiques%204.pdf Le syndrome tardif aux neuroleptiques : quelle place pour la tétrabénazine ?